CLINICAL TRIAL: NCT03015753
Title: A Pilot Randomized Controlled Trial to Test the Complementary Therapeutic Efficacy of Tai Chi for the Prophylaxis of Episodic Migraine in Chinese Women
Brief Title: The Efficacy of Tai Chi Training for the Prophylaxis of Migraine in Chinese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-UA8P
Record Dates: First submitted 2016-12-23; First posted 2017-01-10 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Migraine Disorder
Keywords: Migraine; Tai Chi; Prophylaxis; Randomized controlled trial
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi training (Experimental): The participants in this arm will receive 12-week Tai Chi training (1 hour per day, 5 days per week).
  Interventions: Behavioral: Tai Chi training
- Waiting list control group (Other): Participants in this arm will be asked to maintain their usual lifestyles and exercises for 12 weeks. At the end of the trial , the participants will be offered Tai Chi training similar as Tai Chi group.
  Interventions: Other: Waiting list control group

INTERVENTIONS:
Behavioral: Tai Chi training — The 12-week Tai Chi training will be prescribed with three 1-hour instructor-led sessions and two 1-hour self-practice sessions per week. A modified 32-short form Yang-style Tai Chi Chuan will be adopted. The instructor-led sessions will be operated by qualified Tai Chi masters. The training activity will be delivered in group. The group size is 15 to 18 persons.
  Arms: Tai Chi training
Other: Waiting list control group — At the end of the trial, participants in this arm will be offered Tai Chi training similar as Tai Chi training (TC) group.
  Arms: Waiting list control group

SUMMARY:
The proposed study aims to preliminarily test the effects of a 12-week Tai Chi training on the prophylaxis of episodic migraine in Chinese women, and to evaluate the feasibility, acceptability, compliance and maintenance of Tai Chi exercise among this population.

DETAILED DESCRIPTION:
Migraine is a disabling neurological condition, characterized by attacks of headache and associated symptoms such as photophobia, nausea, and vomiting. In Hong Kong, the overall prevalence is around 12.5%. People with repeated migraine attacks are pain and personal suffering, have impaired social and personal life, and increased financial cost of medication. More nonpharmacologic prophylactic treatments are needed to reduce the high disease burden. As a body-mind exercise, Tai Chi's potential therapeutic efficacy on the prophylaxis of migraine has caught our attention. The investigators propose to conduct a two-arm individual level randomized controlled trial. Local women diagnosed with episodic migraine between 18-65 years will be randomly assigned to one of two groups: 1) a Tai Chi training ("TC"); or 2) a waiting list control group ("control"). The control group will receive a "delayed" Tai Chi training at the end of the trial. A total of 60 participants will be randomized and the intervention period will be 12 weeks with another 12-week follow-up. Number of attacks per month (frequency of attack), intensity and duration of headache, stress, sleep quality and quantity, fatigue, HRQoL, and body composition will be measured at baseline and at 12 weeks and 24 weeks. The primary outcomes are the difference in frequency of attack from baseline to the 12 weeks after randomization, and the proportion of patients with at least a 50% reduction of the number of attacks per month. The intervention effect will be estimated by calculating the differences of outcomes from baseline to the end of the trial between the intervention and control groups using intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-65 years;
* Have a clinical diagnosis of episodic migraine according to ICHD-II criteria at least 2 months prior to enrollment;
* At least one of the following migraine characteristics is met: nausea, vomiting, photophobia, or phonophobia;
* Able to undertake designated level of Tai Chi exercise;
* Live in Hong Kong, can read and speak Cantonese or Putonghua.

Exclusion Criteria:

* Severe migraine attacks with disabilities that cannot perform moderate intensity physical activity;
* Secondary headache and other neurological disease;
* More than 5 days of non-migrainous headache per month;
* Experience with Tai Chi practice after diagnosis of migraine;
* Regular performance of Tai Chi or other body-mind exercises (yoga, biofeedback, medication, etc.);
* Undergoing other alternative therapeutic treatments during recruitment period, or received other alternative therapeutic treatments in the past 12 weeks;
* Pregnancy, lactation period, or currently using contraceptives;
* Use of pharmacological prophylactic treatment for migraine in the past 12 weeks;
* Drug abuse, take antipsychotic or antidepressant drugs, or take analgesics for other chronic pain more than 3 days a month in the past 12 weeks;
* Epilepsy, or have a psychiatric disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The difference in frequency of migraine attacks (the number of attacks per month) | From baseline to 12 weeks
The proportion of responders | From baseline to 12 weeks
  Defined as the proportion of patients with at least a 50% reduction of the number of attacks per month

SECONDARY OUTCOMES:
Duration of headache attack | From the baseline to 12 weeks and 24 weeks
Intensity of headache | From the baseline to 12 weeks and 24 weeks
  Intensity of headache will be measured by a Visual Analogue Scale.
Stress status | From the baseline to 12 weeks and 24 weeks
  The Perceived Stress Scale (PSS) will be used to measure the stress level.
Sleep quality | From the baseline to 12 weeks and 24 weeks
  The Chinese version of the Pittsburgh Sleep Quality Index (PSQI) will be used to measure the sleep quality.
Sleep quantity | From the baseline to 12 weeks and 24 weeks
  A 7-day daily sleep log will be used to measure the sleep quantity.
Fatigue level | From the baseline to 12 weeks and 24 weeks
  The Numeric Rating Scale-fatigue (NRS-fatigue) will be used to measure fatigue level.
HRQoL | From the baseline to 12 weeks and 24 weeks
  HRQoL will be measured by using the Chinese version of the SF-36.
Weight | From the baseline to 12 weeks and 24 weeks
  Weight in kilograms
Height | From the baseline to 12 weeks and 24 weeks
  Height in meters
Waist circumference | From the baseline to 12 weeks and 24 weeks
  Waist in cm
Hip circumference | From baseline to 12 weeks and 24 weeks
  Hip circumference in cm
Percent body fat | From the baseline to 12 weeks and 24 weeks
Session attendance rate | From baseline to 12 weeks
  Number of participants who truly attend the Tai Chi training session divided by the total number of participants in that training session
The number of weeks the participants in intervention group practice Tai Chi at least one time per week in the 12-week follow up period | 12 weeks after Tai Chi training
  This is to measure the maintenance of Tai Chi practice
The percentage of the participants in the intervention group who keep Tai Chi exercise for 1 time per week and last 6 weeks in the 12-week follow up period | 12 weeks after Tai Chi training
  This is to measure the maintenance of Tai Chi practice
Participation rate | At baseline assessment (4 weeks)
  This outcome is measured by the eligible participants at baseline assessment divided by the subjects who register the study
Dropout rate | From the baseline to 12 weeks and 24 weeks
  Number of participants successfully complete the 12-week Tai Chi training and 12-week follow up divided by the number of participants at baseline
Adverse events | During intervention period (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie YJ, Tian L, Hui SS, Qin J, Gao Y, Zhang D, Ma T, Suen LKP, Wang HH, Liu ZM, Hao C, Yang L, Loke AY. Efficacy and feasibility of a 12-week Tai Chi training for the prophylaxis of episodic migraine in Hong Kong Chinese women: A randomized controlled trial. Front Public Health. 2022 Dec 13;10:1000594. doi: 10.3389/fpubh.2022.1000594. eCollection 2022. PMID 36582390
- [Derived] Wang S, Tian L, Ma T, Wong YT, Yan LJ, Gao Y, Zhang D, Hui SS, Xie YJ. Effectiveness of Tai Chi on Blood Pressure, Stress, Fatigue, and Sleep Quality among Chinese Women with Episodic Migraine: A Randomised Controlled Trial. Evid Based Complement Alternat Med. 2022 Oct 19;2022:2089139. doi: 10.1155/2022/2089139. eCollection 2022. PMID 36310622